CLINICAL TRIAL: NCT00006383
Title: Pivotal Phase II Multicenter Study of Vincristine Sulfate Liposomes Injection in Diffuse Large B-Cell Non-Hodgkin's Lymphoma That is Refractory or Relapsed After Second-Line Combination Chemotherapy Revised Title Per 03/01 SR Pivotal Phase II Multicenter Study of Vincristine Sulfate Liposomes Injection in Aggressive Non-Hodgkin's Lymphoma That is Refractory to or Relapsed After Second-Line Combination Chemotherapy
Brief Title: Liposomal Vincristine in Treating Patients With Refractory or Relapsed Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inex Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068259; INEX-CA99002; UCLA-0002028
Record Dates: First submitted 2000-10-04; First posted 2003-05-30 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2002-12

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult T-cell leukemia/lymphoma; anaplastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic

INTERVENTIONS:
Drug: liposomal vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of liposomal vincristine in treating patients who have refractory or relapsed non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the complete and partial tumor responses in patients with aggressive non-Hodgkin's lymphoma that is refractory to or relapsed after second-line combination chemotherapy treated with vincristine sulfate liposomes injection.
* Determine the toxicity of this treatment regimen in these patients.
* Determine the duration of response, time to progression, and survival in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive vincristine sulfate liposomes IV over 1 hour. Treatment repeats every 2 weeks for a maximum of 12 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 8 weeks until disease progression.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed aggressive non-Hodgkin's lymphoma including:

  * Peripheral T-cell lymphoma not otherwise specified
  * Anaplastic large null-/T-cell lymphoma
  * Diffuse large B-cell lymphoma including:

    * Primary mediastinal large B-cell lymphoma with sclerosis
    * Intravascular large B-cell lymphoma
    * Immunoblastic B-cell lymphoma
    * T-cell-rich B-cell lymphoma
    * Anaplastic large B-cell lymphoma
* At least one bidimensionally measurable lesion with clearly defined margins at least 2 cm in the largest dimension by physical examination or CT scan
* No prior or active CNS lymphoma or AIDS-related lymphoma
* Must have received 2 or more prior chemotherapy courses from time of diagnosis of aggressive lymphoma or from time of biopsy-proven transformation from indolent to aggressive

  * Prior first and second-line therapy must have been combination chemotherapy
  * Prior first-line chemotherapy regimen must have contained anthracycline
  * Must have had at least a minor response to first-line therapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-3

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 500/mm^3 (unless due to lymphoma bone marrow involvement)
* Platelet count at least 50,000/mm^3 (unless due to lymphoma bone marrow involvement)

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* ALT no greater than 4 times ULN
* Alkaline phosphatase no greater than 4 times ULN

Renal:

* Not specified

Neurologic:

* No prior neurological disorders unrelated to chemotherapy (including familial neurological diseases or acquired demyelinating disorders)
* No neuromuscular impairment (neuromotor, neurosensory, or neurocerebellar)
* No prior grade 3 or 4 sensory or motor neuropathy related to chemotherapy

Other:

* No uncontrolled severe medical illness or infection
* HIV negative
* No other malignancies within the past 5 years except curatively resected basal cell skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Radiotherapy
* No prior allogeneic bone marrow or peripheral blood stem cell transplantation
* At least 4 weeks since prior immunotherapy
* No concurrent biological agents

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* At least 4 weeks since prior corticosteroids at a dose greater than 10 mg/day of prednisone or equivalent

Radiotherapy:

* Prior involved-field radiotherapy allowed if irradiated area is not the only source of measurable disease
* Prior total body radiotherapy with high-dose therapy and autologous stem cell transplantation allowed
* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy to any disease site

Surgery:

* At least 4 weeks since prior major surgery except for diagnosis of lymphoma
* No concurrent surgical removal of any indicator lesion

Other:

* At least 4 weeks since prior alternative or investigational anticancer treatment
* No other concurrent systemic anticancer therapy
* No other concurrent investigational drug
* No concurrent phenytoin
* No concurrent hepatic drug metabolism inhibitors or inducers (cytochrome P450 isoenzymes in the CYP 3A subfamily)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06; Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gallimore, PhD, Study Chair — Inex Pharmaceuticals
Locations (9):
- United States (8):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - University of Texas Health Center at Tyler, Tyler, Texas
  - Vermont Cancer Center, Burlington, Vermont
- Tom Baker Cancer Center - Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Result] Rodriguez MA, Pytlik R, Kozak T, Chhanabhai M, Gascoyne R, Lu B, Deitcher SR, Winter JN; Marqibo Investigators. Vincristine sulfate liposomes injection (Marqibo) in heavily pretreated patients with refractory aggressive non-Hodgkin lymphoma: report of the pivotal phase 2 study. Cancer. 2009 Aug 1;115(15):3475-82. doi: 10.1002/cncr.24359. PMID 19536896